CLINICAL TRIAL: NCT01542775
Title: Effects of Exercise on sRAGE Levels and Cardiometabolic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Clinical Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Exer(sRAGE)
Record Dates: First submitted 2012-02-20; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Control Groups

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Behavioral: Control Group
- Exercise (Active Comparator)
  Interventions: Behavioral: Aerobic Exercise Group

INTERVENTIONS:
Behavioral: Aerobic Exercise Group — 12 weeks Aerobic exercise
  Arms: Exercise
Behavioral: Control Group — maintaining usual activities
  Arms: Control

SUMMARY:
The purpose of this study is to examine the effects of exercise on diverse cardiometabolic risk factors and indicators of atherosclerosis in patients with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* stable body weight
* sedentary lifestyle

Exclusion Criteria:

* smoked cigarettes
* cardiovascular disease
* chronic kidney
* chronic liver disease
* pregnant or breastfeeding
* any other major illness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change from baseline in soluble receptor for advanced glycation endproducts (sRAGE) after 12 weeks of aerobic exercise | 12 weeks

SECONDARY OUTCOMES:
anthropometric parameters | 12 weeks
  body weight, waist circumference, body fat percentage, visceral fat area
biochemical parameters | 12 weeks
  HbA1c, apolipoprotein B, free fatty acid
energy expenditure | 12 weeks
  activity energy expenditure, total energy expenditure

CONTACTS AND LOCATIONS:
Locations (1):
- Eulji University School of Medicine, Seoul, South Korea